CLINICAL TRIAL: NCT03791827
Title: Multicenter Registry of Pediatric Lupus Nephritis in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiqiang Dang (Other)
Collaborators: The Children's Hospital Affiliated to Suzhou University (Unknown); Shandong Provincial Hospital (Other Government); Guizhou Provincial People's Hospital (Other); LanZhou University (Other); The First Affiliated Hospital of Inner Mongolia Medical College (Unknown); People's Hospital of Zhangjiajie (Unknown); Puyang Oilfield General Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Guizhou Maternal and Child Health Care Hospital (Unknown); The Second Affiliated Hospital & Yuying Children's Hospital of Wenzhou Medical University (Unknown); Shenzhen Children's Hospital (Other Government); The Second Affiliated Hospital of Harbin Medical University (Other); Yichang Central People's Hospital (Other); Xian Children's Hospital (Other Government); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The First People's Hospital of Yunnan (Other); The First Affiliated Hospital of Xiamen University (Other); The First Affiliated Hospital of Xinxiang Medical College (Other); Shanxi Provincial Maternity and Children's Hospital (Other); Liaocheng People's Hospital (Other); Fujian Provincial Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Lanzhou University Second Hospital (Other); Guangzhou First People's Hospital (Other); The Second Hospital of Shandong University (Other); Children's Hospital of Hebei Province (Other); Beijing Children's Hospital (Other); Zhengzhou Children's Hospital (Unknown); The Children's Hospital of Chongqing Medical University (Unknown); Wuxi Women's & Children's Hospital (Other); The Children's Hospital of Fudan University (Unknown); Shanghai Children's Medical Center (Other); Qilu Children's Hospital of Shandong University (Other)
Responsible Party: Sponsor-Investigator, Xiqiang Dang, Professor, Second Xiangya Hospital of Central South University
Organization: Second Xiangya Hospital of Central South University (Other)
Other Study IDs: Pediatric lupus nephritis
Record Dates: First submitted 2018-12-24; First posted 2019-01-03 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Lupus Nephritis; Children; Steroid; Immunosuppressive Treatment
MeSH Terms: conditions — Lupus Nephritis | interventions — Adrenal Cortex Hormones; Steroids; Prednisone; Prednisolone; Hydroxychloroquine; Cyclophosphamide; Mycophenolic Acid; Azathioprine; Tacrolimus; Cyclosporine; Rituximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (8):
- Corticosteroid: Pediatric lupus nephritis treated with hydroxychloroquine and corticosteroid
  Interventions: Drug: Corticosteroid; Drug: Hydroxychloroquine
- Corticosteroid and cyclophosphamide: Pediatric lupus nephritis treated with hydroxychloroquine, corticosteroid and cyclophosphamide
  Interventions: Drug: Corticosteroid; Drug: Hydroxychloroquine; Drug: Cyclophosphamide
- Corticosteroid and mycophenolate mofetil: Pediatric lupus nephritis treated with hydroxychloroquine, corticosteroid and mycophenolate mofetil
  Interventions: Drug: Corticosteroid; Drug: Hydroxychloroquine; Drug: Mycophenolate Mofetil
- Corticosteroid and azathioprine: Pediatric lupus nephritis treated with hydroxychloroquine, corticosteroid and azathioprine
  Interventions: Drug: Corticosteroid; Drug: Hydroxychloroquine; Drug: Azathioprine
- Corticosteroid and tacrolimus: Pediatric lupus nephritis treated with hydroxychloroquine, corticosteroid and tacrolimus
  Interventions: Drug: Corticosteroid; Drug: Hydroxychloroquine; Drug: Tacrolimus
- Corticosteroid and cyclosporine A: Pediatric lupus nephritis treated with hydroxychloroquine, corticosteroid and cyclosporine A
  Interventions: Drug: Corticosteroid; Drug: Hydroxychloroquine; Drug: Cyclosporine A
- Corticosteroid, mycophenolate mofetil and tacrolimus: Pediatric lupus nephritis treated with hydroxychloroquine, corticosteroid, mycophenolate mofetil and tacrolimus
  Interventions: Drug: Corticosteroid; Drug: Hydroxychloroquine; Drug: Azathioprine; Drug: Cyclosporine A
- Retuximab: An option for refractory lupus nephritis
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Corticosteroid — corticosteroid is given to patients orally or methylprednisone is given to patients through i.v.
  Other Names: Steroid; Prednisone; Methylprednisone; Prednisolone
  Groups: Corticosteroid; Corticosteroid and azathioprine; Corticosteroid and cyclophosphamide; Corticosteroid and cyclosporine A; Corticosteroid and mycophenolate mofetil; Corticosteroid and tacrolimus; Corticosteroid, mycophenolate mofetil and tacrolimus
Drug: Hydroxychloroquine — Hydroxychloroquine is recommended as the basic therapy for lupus nephritis
  Groups: Corticosteroid; Corticosteroid and azathioprine; Corticosteroid and cyclophosphamide; Corticosteroid and cyclosporine A; Corticosteroid and mycophenolate mofetil; Corticosteroid and tacrolimus; Corticosteroid, mycophenolate mofetil and tacrolimus
Drug: Cyclophosphamide — The typical therapy for cyclophosphamide is either 500 to 750mg/m2 once every month for 6 doses or 8 to 12 mg/kg/d for two consecutive days every two weeks for 6 to 8 doses through i.v.
  Groups: Corticosteroid and cyclophosphamide
Drug: Mycophenolate Mofetil — The recommended dose of mycophenolate mofetil is 20 to 30mg/kg/d
  Groups: Corticosteroid and mycophenolate mofetil
Drug: Azathioprine — The recommended dose of azathioprine is 1.5 to 2mg/kg/d
  Groups: Corticosteroid and azathioprine; Corticosteroid, mycophenolate mofetil and tacrolimus
Drug: Tacrolimus — The recommended dose of tacrolimus is 0.05 to 0.15mg/kg/d, Q12h
  Groups: Corticosteroid and tacrolimus
Drug: Cyclosporine A — The recommended initial dose of cyclosporine A is 4 to 6mg/kg/d, Q12h
  Groups: Corticosteroid and cyclosporine A; Corticosteroid, mycophenolate mofetil and tacrolimus
Drug: Rituximab — The recommended dose of rituximab is 375mg/m2 once a week for 2 to 4 doses
  Other Names: anti-CD20 antibody
  Groups: Retuximab

SUMMARY:
This study is designed to evaluate the efficacy and safety of the current treatment option and outcome of pediatric lupus nephritis patients in China. Investigators will perform prospective registration study among at least 35 pediatric nephrology medical centers in China.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of lupus nephritis:

* Diagnosis of SLE according to the 1997 update of the 1982 American College of Rheumatology revised criteria for classification of systemic lupus erythematosus
* Either of the following: Positive urine protein detected 3 times within a week, or 24-hour urine protein>150mg, or UPC>0.2mg/mg, or urinary microalbumin above normal range detected 3 times within a week, or microscopic examination erythrocyte>5 RBC/HP, or renal dysfunction including glomerular and/or tubular dyfunction, or abnormal renal biopsy and the pathological changes are in accordance with lupus nephritis
* The pathological diagnosis of kidney conforms to the International Society of Nephrology and Society of Renal Pathology (ISN/RPS) standards in 2003

Exclusion Criteria (either of the following criteria):

* Complicated with other systemic diseases, including basic diseases with clinical significance
* Patients with tumors
* Patients with abnormal glucose metabolism
* Immunodeficiency patients
* Patients diagnosed as tuberculosis, or hepatitis B, or hepatitis C within three months before treatment
* Patients with other connective tissue diseases (such as Sjogren's syndrome, mixed connective tissue disease, etc.)
* Drug-induced lupus, congenital lupus and other secondary lupus
* Renal histopathology with non-inflammatory necrotizing angiopathy or thrombotic microangiopathy (TMA)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 1200 pediatric lupus nephritis patients younger than 18 years old will be enrolled from more than 35 pediatric nephrology medical centers nationwide
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Complete remission | 5 years
  complete remission is defined as UPC<0.2 mg/mg， or 24-hour urine protein<150mg with normal kidney function and without hematuria
Partial remission | 5 years
  Partial remission is defined as non-nephrotic range proteinura, decrease of urine protein ≥50%， and serum creatinine remains stable (±25% of baseline) or is improved but not normal yet

SECONDARY OUTCOMES:
End stage renal disease (ESRD) | 1 year, 2 years, 3 years, 4 years and 5 years
  ESRD is defined as eGFR<15ml/1.73m2, initiation of long-term dialysis or kidney
Mortality | 1 year, 2 years, 3 years, 4 years and 5 years
  Death of patients

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
Currently, IPD is not available to other researchers